CLINICAL TRIAL: NCT06748144
Title: Intraosseous vs. Intravenous Vancomycin Administration in Spine Surgery
Brief Title: IO Vancomycin Spine
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Mark Prasarn, Orthopedic Surgeon, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00038766
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Fusion Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous Vancomycin (Experimental): Participants in this group will receive other antibiotics according to the Houston Methodist Hospital orthopedic surgeon's standard of care regimen, which typically involves ancef or cefepime being administered in pre-op within 1 hour of the incision. IO Vancomycin will be administered in the OR after incision (500mg in 100-150mL normal saline (NS)), and the injection will be placed into the posterior ilium.
  Interventions: Drug: Intraosseous Vancomycin
- Intravenous Vancomycin (Active Comparator): Patients will receive the Houston Methodist Hospital orthopedic surgeon's standard of care pre-operative antibiotic regimen for lumbar fusion patients. This includes IV antibiotics (typically ancef or cefepime and vancomycin), which will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg, generally 1000-1750mg in 500mL NS).
  Interventions: Drug: Intravenous Vancomycin

INTERVENTIONS:
Drug: Intraosseous Vancomycin — The intervention is specific to the method of administration that will be used when giving the dose of antibiotic vancomycin which is done to prevent infection following surgery.
  Arms: Intraosseous Vancomycin
Drug: Intravenous Vancomycin — This is the standard method of giving the antibiotic vancomycin to patients undergoing surgery across many specialties in order to prevent infection.
  Arms: Intravenous Vancomycin

SUMMARY:
The goal of this research is to learn if injecting the antibiotic vancomycin directly into the bone marrow (intraosseous) or IO) during a lumbar (spinal) fusion surgery, is as effective or better than the standard method of giving it vancomycin through a vein (intravenous) or IV) during lumbar fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing open posterior instrumented spinal fusion (PSIF) or transforaminal lumbar interbody fusion (TLIF)
* Patient is able to give informed consent to participate on the study. LAR consents will not be utilized for this study
* Age Range >18

Exclusion Criteria:

* Previous spine surgery if surgeon deems it will affect the study
* BMI > 40
* Contraindication to receiving vancomycin, cefepime, ancef, or other standard of care pre-operative antibiotic (allergy, medical issue, etc).
* Inability to administer the IO infusion
* Refusal to participate
* Diabetes as defined as uncontrolled A1C > 7.5 and eGFR <59
* Immunocompromised or immunosuppressed patients (HIV, Hep C, ESRD, dialysis, transplant, chemo/radiation treatment in last 6 months, medications)
* No vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Change in Level of Systemic Vancomycin Concentration | Start of skin incision during surgery, Start of closure of skin incision during surgery
  The level of vancomycin concentration will be assessed via a blood draw by the anesthesiologist staff.
Level of Vancomycin Concentration in Bone | During surgery
  Bony tissue samples (Superior Articular Process, Inferior Articular Process, and Lamina) will be taken during surgery to assess levels of vancomycin concentration in the bone.
Level of Vancomycin Concentration in Soft Tissue | During surgery
  Soft tissue samples (Multifidus muscle, Fat) will be taken during surgery to assess levels of vancomycin concentration in the tissue.

SECONDARY OUTCOMES:
Post-Operative Complication Rates | 30 Days Post Surgery, 90 Days Post Surgery
  Participant's charts will be reviewed postoperatively to determine if there were any adverse local/systemic reactions and/or complications following the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No